CLINICAL TRIAL: NCT01079650
Title: Diagnosis of Acute Appendicitis, Ovary Torsion and Inflammation, and Testicular Torsion and Inflammation by Infrared Thermography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Diagnosis of acute appendicitis, ovary torsion and inflammation, and testicular torsion and inflammation by infrared thermography., Assaf-Harofeh Medical Center, Anesthesiology department.
Other Study IDs: 39/10
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Abdominal Pain; Testicle Pain
Keywords: children
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- children suffering from abdominal or testicle pain

SUMMARY:
Thermal, or infrared, energy is the part of electromagnetic radiation that an observer perceives as heat. Infrared thermography allows us to visualize temperature distribution of the human body and has been used in medical practice since the 1950s. In current study we would like to examine the ability of infrared thermography to detect acute appendicitis, ovary torsion and inflammation, and testicular torsion and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years old

Exclusion Criteria:

* > 18 years old

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children (<18 years old) having abdominal or testicle pain.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh MC, Beer-Yaakov, Israel